CLINICAL TRIAL: NCT00490880
Title: The Evaluation of Efficacy and Toxicity of Combined Treatment: Neoadjuvant Chemotherapy (Gemcitabine and Cisplatin) With Radical Cystectomy or Radiotherapy in Patients With Bladder Cancer Stage T2b-T3 NO/Nx M0
Brief Title: Neoadjuvant Chemo (Gemcitabine and Cisplatin) With Radical Cystectomy or Radiotherapy in Patients With Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8193; B9E-MC-S341
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Cisplatin; Cystectomy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: gemcitabine
Drug: cisplatin
Procedure: radical cystectomy
Procedure: radiotherapy

SUMMARY:
The purpose of this study is to evaluate efficacy of gemcitabine and cisplatin combined with either radical cystectomy or radiotherapy in the treatment of bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven urothelial carcinoma of the urinary bladder in stage T2b-T3, N0/Nx, M0.
* Patients must have measurable disease. Response assessment will be evaluated according to RECIST criteria. Measurable lesions with clearly defined margins will be evaluated by X-Ray, Transvesical Ultrasound, CT-Scan or MRI, cystoscopy.
* Lesions serving as measurable disease must have the longest diameter of greater than or equal to 20 mm as measured with conventional techniques or greater than or equal 10 mm with spiral CT scan. Lesions measured by physical examination must have a longest diameter of greater than or equal 20 mm.

Exclusion Criteria:

* Patients with prior or concomitant malignant diseases (other than appropriately treated basal cell carcinoma of the skin or carcinoma of the cervix)
* PSA greater than 5.0 ng/mL
* Concurrent administration of any other tumor therapy, including radiotherapy, cytotoxic chemotherapy, immunotherapy, molecular target therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2003-11; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
To evaluate efficacy

SECONDARY OUTCOMES:
To evaluate pathological complete responses
To evaluate progression free survival
To evaluate overall survival
To evaluate time to disease progression
To evaluate safety

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw, Poland

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com